CLINICAL TRIAL: NCT06760013
Title: The Effect of Su-jok Therapy Applied in the First Stage of Labor on Pain Level in Primiparas
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, AYSUDA REFİYE AKVERAN, Graduate Student, Hitit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HU-SBF-ARA-01
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Labor Pain
Keywords: su jok therapy; labor pain; primiparous
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: It is planned to have a Randomized Control experimental design in two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Su jok therapy group (Active Comparator): Sujok massage therapy will be applied to the affected area on the hands of pregnant women who will give birth for the first time.
  Interventions: Behavioral: Su Jok Therapy
- Control Group (No Intervention): A comparison will be made on this group with pregnant women who receive sujok therapy without any therapy.

INTERVENTIONS:
Behavioral: Su Jok Therapy — The researcher, who has a Su-Jok practitioner certificate, applied pressure for 1-2 minutes on the active point on the meridian (the area between the 3rd and 4th fingers pointing to the uterus) that provides energy flow in the palm in 20-minute periods, with the help of a diagnostic probe (diagnostic stick). The point will be determined. Once this point is detected, a massage will be performed on the point. The massage will be applied with a 10-minute rest period between each two periods.
  Arms: Su jok therapy group

SUMMARY:
The aim of this study is to examine the effect of sujok therapy applied in the first stage of labor on the pain level in primiparas.

DETAILED DESCRIPTION:
Birth pain, known as acute pain, is felt in the human body as one of the oldest, complex, severe and most difficult to control types of pain. However, this pain differs from other types of pain due to the fact that it reunites the mother with her baby and covers a limited period of time. Pain is a subjective phenomenon that every individual experiences throughout their lives and to which people react differently.

Su Jok therapy, an alternative and complementary therapy technique, is seen as a method that balances the energy flow based on the philosophy of non-pharmacological and non-invasive acupuncture that can be used to control labor pain.

Su-jok application is the development of a massage therapy that will create a feeling of comfort in the body by using certain points. There are tiny swellings on the reflection points on the hands and feet (such as the area between the 3rd and 4th fingers reflecting the uterus area). These are also called micro acupuncture points. When pressure is applied to these swellings on the hands and feet for 1-2 minutes, pain and a feeling of pulling occur. Thus, the area to be massaged is determined. During the detection phase, a blunt-tipped diagnostic probe or a round-tipped stick can be used. At this stage, the same amount of pressure should be applied to the area to be applied. When a point is determined, the correct point for massage application should be massaged and energy flow should be provided. Since it does not have any side effects, it is a therapy that can be used in pregnant women and is a massage application that does not require any invasive intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being primiparous
* The pregnant woman must be over 18 years of age
* To participate in the research voluntarily
* The beginning of labor (water breaking, presence of non-stress testa contractions, engagement)

Exclusion Criteria:

* Pregnancies outside 37-41 weeks
* Multiparas
* Those who are not pregnant
* Having visual, mental and auditory disabilities
* Being pregnant as an adolescent
* Not accepting participation in the research

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since the therapy method to be applied is performed on pregnant women, it will only be applied to women.
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | eight months
  A number indicating the pain level will be expressed on the scale between 1-10.

SECONDARY OUTCOMES:
MONITORING FORM FOR BIRTH (FOR SU JOK GROUP) | eight months
  It is a survey that includes pregnant women's information about birth and their opinions on su jok therapy.
MONITORING FORM FOR BIRTH (CONTROL GROUP) | eight months
  The survey, which consists of nine questions, includes information about the birth process of pregnant women. (Vitals, vaginal examination findings)

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University, Çorum, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No